CLINICAL TRIAL: NCT04043845
Title: A Phase 1 Study Targeting ERK 1/2 Signaling in Ibrutinib Resistant B-cell Malignancies
Brief Title: ERK 1/2 Signaling in Ibrutinib Resistant B-cell Malignancies
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Business development reasons.
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Principal Investigator, Steven P. Treon, MD, PhD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19-277
Record Dates: First submitted 2019-07-31; First posted 2019-08-02 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-02

CONDITIONS: Chronic Lymphocytic Leukemia; Waldenstrom Macroglobulinemia; Mantle Cell Lymphoma; Marginal Zone Lymphoma
Keywords: Chronic Lymphocytic Leukemia; Waldenstrom Macroglobulinemia; Mantle Cell Lymphoma; Marginal Zone Lymphoma; CLL; WM; MCL; MZL; ERK; Ibrutinib; BTKCys481; PLCG2; PLCγ2; LY3214996
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Waldenstrom Macroglobulinemia; Lymphoma, Mantle-Cell; Lymphoma, B-Cell, Marginal Zone | interventions — ibrutinib; LY3214996

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- LY3214996+Ibrutinib (Experimental): * LY3214996 will be administered by mouth once daily continuously throughout each treatment cycle
  * Ibrutinib will be administered by mouth once daily continuously throughout each treatment cycle.
  Interventions: Drug: Ibrutinib; Drug: LY3214996

INTERVENTIONS:
Drug: Ibrutinib — Ibrutinib inhibits the function of Bruton's tyrosine kinase (BTK). Ibrutinib blocks signals that stimulate malignant B cells to grow and divide uncontrollably.
  Other Names: Imbruvica
Drug: LY3214996 — LY3214996 is an extracellular signal-regulated kinase (ERK) inhibitor. ERK inhibitors stop the signal that a cancer cell receives telling it to grow.

SUMMARY:
This research is studying the safety of combining ibrutinib with the study drug LY3214996 for chronic lymphocytic leukemia (CLL), Waldenstrom's macroglobulinemia (WM), mantle cell lymphoma (MCL), or marginal zone lymphoma (MZL).

DETAILED DESCRIPTION:
This research study is a Phase I clinical trial, which tests the safety of an investigational combination of drugs and also tries to define the appropriate dose of the investigational drug to use for further studies. "Investigational" means that the drug is being studied.

The U.S. Food and Drug Administration (FDA) has not approved LY3214996 as a treatment for any disease.

The U.S. Food and Drug Administration (FDA) has approved ibrutinib as a treatment option for this disease.

LY3214996 is an extracellular signal-regulated kinase (ERK) inhibitor that is being developed as a treatment for patients with advanced cancer. ERK inhibitors stop the signal that a cancer cell receives telling it to grow. In this research study, the investigators are testing to see if LY3214996 is safe when combined with ibrutinib in patients with specific gene mutations. Making treatment decisions based on genetic testing is investigational, and the FDA has not approved this genetic testing. Several doses of LY3214996 will be explored in this study.

ELIGIBILITY:
Inclusion Criteria:

* Participants must meet one of the following criteria:

  * Clinicopathological diagnosis of Waldenstrom's macroglobulinemia (WM) meeting criteria for treatment using consensus panel guidelines from the Second International Workshop on Waldenstrom's Macroglobulinemia31 or have high risk disease with a serum IgM level of 6,000 mg or higher.32
  * Confirmed diagnosis of chronic lymphocytic leukemia (CLL) per International Workshop on CLL 2018 criteria.33
  * Histologically or cytologically confirmed diagnosis of mantle cell lymphoma (MCL) or marginal zone lymphoma (MZL).
* Participants must have a BTKCys481 and/or PLCγ2 mutation. Genomic alterations must have been confirmed via sequencing performed at NeoGenomics Laboratories.
* All participants must have experienced disease progression while actively receiving ibrutinib monotherapy based on National Comprehensive Cancer Network (NCCN) guidelines.
* All participants must be actively receiving ibrutinib monotherapy at the time of study entry. Participants with a gap in treatment or who received anti-cancer treatments other than ibrutinib immediately prior to study entry are not eligible.
* Participants must have been on a stable dose of ibrutinib monotherapy for a minimum of 3 weeks prior to cycle 1 day 1.
* Age ≥ 18 years.
* ECOG performance status ≤ 1 (see Appendix A)
* Participants must have measurable disease:

  * Participants with WM: presence of serum immunoglobulin M (IgM) with a minimum IgM level of > 2 × institutional upper limit of normal.
  * Participants with CLL:

    * Palpable or CT measurable lymphadenopathy ≥ 1.5 cm, AND/OR
    * Lymphocytosis ≥ 5,000/μL, AND/OR
    * Bone marrow involvement of ≥ 30%
  * Participants with MCL or MZL: at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded for non-nodal lesions and short axis for nodal lesions) as ≥ 20 mm (≥ 2 cm) with conventional imaging or > 10 mm with spiral CT scan. If the patient has been previously irradiated, there must be evidence of progression in the lesion since the radiation.
* Participants must have adequate organ and marrow function as defined below:

  * Absolute Neutrophil Count ≥ 750/mcL
  * Platelet Count ≥ 50,000/mcL
  * Total Bilirubin ≤ 1.5 × institutional upper limit of normal (ULN), OR
  * Total Bilirubin ≤ 2 × institutional ULN if elevation is attributable to Gilbert's syndrome
  * AST (SGOT) / ALT(SGPT) ≤ 2.5 × institutional ULN, OR
  * AST (SGOT) / ALT (SGPT) ≤ 5 × institutional ULN if elevation is a result of infiltration by neoplastic disease
  * Creatinine ≤ 1.5 × institutional ULN, OR
  * Creatinine Clearance ≥ 60 mL/min/1.73 m2 for participants with creatinine levels above 1.5 × institutional normal (calculated via the Cockcroft-Gault equation)
* The effects of ibrutinib or LY3214996 on the developing human fetus are unknown. For this reason and because anti-cancer agents are known to be teratogenic, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 4 months after completion of ibrutinib or LY3214996 administration.
* Ability to understand and the willingness to sign a written informed consent document.
* Ability to swallow and retain oral medication.

Exclusion Criteria:

* Participants who have had major surgery within 4 weeks prior to the first dose of study medication.
* Participants who have previously received treatment with an ERK inhibitor, including but not limited to previous treatment with LY3214996.
* Participants with known CNS disease involvement should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to LY3214996 or ibrutinib.
* Individuals with a history of a different malignancy are ineligible with the following exceptions: individuals who have been treated and are disease-free for a minimum of 3 years prior to study enrollment, or individuals who are deemed by the treating investigator to be at low risk for disease recurrence. Additionally, individuals with the following cancers are eligible if diagnosed within the past 3 years: basal or squamous cell carcinomas of the skin, breast or cervical carcinomas in situ, and low risk prostate cancer that does not require treatment as judged by the treating investigator.
* Participants who are known at the time of trial enrollment to require concomitant therapy with strong or moderate CYP3A inhibitors or inducers. The use of strong or moderate CYP3A inhibitors or inducers is prohibited for the duration of trial treatment.
* Participants who are known at the time of trial enrollment to require concomitant therapy with sensitive substrates of CYP3A4 or drugs cleared by CYP3A4 that have a narrow therapeutic range. The use of these drugs is prohibited for the duration of trial treatment.
* Uncontrolled intercurrent illness including, but not limited to: ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant women are excluded from this study because LY3214996 and ibrutinib are agents with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with LY3214996 or ibrutinib, breastfeeding should be discontinued if the mother is treated with LY3214996 or ibrutinib. A negative serum pregnancy test is required for women of childbearing potential prior to the first dose of study medication.
* Participants who are known to be seropositive for human immunodeficiency virus (HIV) or hepatitis B or C.
* Participants with a history or findings of central or branch retinal artery or venous occlusion with significant vision less, or other retinal diseases causing visual impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-02-03 (Actual); Primary Completion 2020-02-03 (Actual); Study Completion 2020-02-03 (Actual)

PRIMARY OUTCOMES:
Dose Limiting Toxicity | 42 days
  Toxicities occurring following administration of protocol therapy, measured using CTCAE 5.0 criteria.

SECONDARY OUTCOMES:
Best Response | From date of study drug initiation up to a maximum of 2 years
  Best response to study treatment measured using disease-specific criteria.
Time to Progression | From date of study drug initiation until the date of first documented progression or date of death from any cause, whichever comes first, up to a maximum of 2 years
  Assess the amount of time to disease progression

CONTACTS AND LOCATIONS:
Overall Officials: Steven Treon, MD, PhD, Principal Investigator — Dana-Farber Cancer Institute

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: BCH - Contact the Technology & Innovation Development Office at www.childrensinnovations.org or email TIDO@childrens.harvard.edu BIDMC - Contact the Beth Israel Deaconess Medical Center Technology Ventures Office at tvo@bidmc.harvard.edu BWH - Contact the Partners Innovations team at http://www.partners.org/innovation DFCI - Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu MGH - Contact the Partners Innovations team at http://www.partners.org/innovation